CLINICAL TRIAL: NCT00850889
Title: Juvederm Ultra With Lidocaine Compared With Restylane for the Correction of Nasolabial Folds
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan Medical (Industry)
Responsible Party: Sponsor
Organization: Allergan (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MA-JULIDO-0801
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Results first posted 2011-04-21 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Nasolabial Folds
Keywords: Aesthetic correction of nasolabial folds

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 1 (Active Comparator): Juvederm Ultra Injectable Gel with Lidocaine
  Interventions: Device: Hyaluronic acid gel (24 mg/mL) with 0.3% lidocaine
- 2 (Active Comparator): Restylane Injectable Gel
  Interventions: Device: A gel of hyaluronic acid (concentration of 20 mg/mL)

INTERVENTIONS:
Device: Hyaluronic acid gel (24 mg/mL) with 0.3% lidocaine — Day 0, maximum total volume (dosage) allowed for each NLF is 1.6 mL
  Other Names: Juvederm® Ultra Injectable Gel with Lidocaine
  Arms: 1
Device: A gel of hyaluronic acid (concentration of 20 mg/mL) — Day 0, maximum total volume (dosage) allowed for each NLF is 1.6 mL
  Other Names: Restylane® Injectable Gel
  Arms: 2

SUMMARY:
Comparison of the safety and effectiveness of Juvederm Ultra with lidocaine compared with Restylane in the correction of nasolabial folds.

ELIGIBILITY:
Inclusion Criteria:

* Desires correction of moderate to severe nasolabial folds (NLFs)
* Both NLFs have the same pre-treatment NLF severity score (either moderate or severe)
* Females of childbearing potential must have a negative urine pregnancy test result at baseline and practice a reliable method of contraception throughout the study

Exclusion Criteria:

* Cosmetic facial procedures [e.g., facelift, resurfacing (laser, photomodulation, intense pulsed light, radio frequency, dermabrasion, chemical peel or other ablative or non-ablative procedures), tissue augmentation with dermal fillers or fat injections, BOTOX Cosmetic injections, or mesotherapy] in the lower 2/3 of the face, including the neck, within 1 month prior to study entry or be planning to undergo any of these procedures at any time during the study
* Initiating use of any new over-the-counter or prescription, oral or topical, anti-wrinkle products in the NLF area within 1 month prior to enrollment or during the study
* Previous hyaluronic acid (HA)-based dermal filler treatment(s) injected within the last 12 months prior to enrollment is within 5mL of the recommended annual maximum volume for HA dermal fillers
* Previous injection of semi-permanent fillers or placement of facial implants anywhere in the head and neck or implantation of any of these products during the study
* Allergy or sensitivity to lidocaine, hyaluronic acid products, or Streptococcal protein
* Active inflammation, infection, cancerous or pre-cancerous lesion or unhealed wound in the NLF region
* Current treatment with anti-coagulation therapy or use of non-steroidal anti-inflammatory drugs or other substances known to increase coagulation time within 10 days of undergoing study injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Niagara Falls, Ontario, Canada

REFERENCES:
- [Background] Smith SR, Jones D, Thomas JA, Murphy DK, Beddingfield FC 3rd. Duration of wrinkle correction following repeat treatment with Juvederm hyaluronic acid fillers. Arch Dermatol Res. 2010 Dec;302(10):757-62. doi: 10.1007/s00403-010-1086-8. Epub 2010 Oct 9. PMID 20936295

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment:32 Study Start Date: November 2008 Study Completion Date: February 2009 Primary Completion Date: November 2008
Groups:
- Total Participants: Each participant received Juvederm on one side of the face and Restylane on the other side.
Period: Overall Study
Arm/Group | Total Participants
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total Participants
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (7.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 1
Region of Enrollment [Number; unit: participants]
  Canada | 32

OUTCOME MEASURES:

1. Primary Outcome: Procedural Pain Score
Description: Subjects evaluated the pain associated with the procedure on an 11-point scale, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Juvederm(R) Ultra Injectable Gel With Lidocaine | Restylane(R) Injectable Gel
Number analyzed (Participants) | 32 | 32
units on a scale | 2.0 (1.84) | 4.1 (1.88)

2. Secondary Outcome: Comparative Pain
Description: A 5-point scale (-2 = Juvéderm with Lidocaine less painful than Restylane; -1 = Juvéderm with Lidocaine slightly less painful than Restylane; 0 = No difference; 1 = Juvéderm with Lidocaine slightly more painful than Restylane; 2 = Juvéderm with Lidocaine more painful than Restylane). Subjects selected one category from the scale; the percentage of subjects that selected each category is presented.
Time Frame: 1 day
Measure: Number; unit: percent of participants
Arm/Group | Total Study Participants
Number analyzed (Participants) | 32
percent of participants
  Juvederm with Lidocaine less painful than Restylan | 34
  Juvederm with Lidocaine slightly less painful than | 50
  No difference | 3
  Juvederm with Lidocaine slightly more painful than | 9
  Juvederm with Lidocaine more painful than Restylan | 3

3. Secondary Outcome: Investigator Assessment of Improvement Since Baseline in Nasolabial Fold (NLF) Severity
Description: Investigator determination of improvement in NLF severity score on 5-point NLF Severity Scale (0 = None; 1 = Mild; 2 = Moderate; 3 = Severe; 4 = Extreme) two weeks after treatment with Juvéderm with Lidocaine in one NLF and Restylane in the other NLF
Time Frame: Day 0, Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Juvederm(R) Ultra Injectable Gel With Lidocaine | Restylane(R) Injectable Gel
Number analyzed (Participants) | 32 | 32
units on a scale | 1.4 (0.91) | 1.3 (0.90)

4. Secondary Outcome: Subject Assessment of Improvement From Baseline in Nasolabial Fold (NLF) Severity
Description: Subject determination of improvement in NLF severity score on 5-point NLF Severity Scale (0 = None; 1 = Mild; 2 = Moderate; 3 = Severe; 4 = Extreme) two weeks after treatment with Juvéderm with Lidocaine in one NLF and Restylane in the other NLF
Time Frame: Day 0, Day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Juvederm(R) Ultra Injectable Gel With Lidocaine | Restylane(R) Injectable Gel
Number analyzed (Participants) | 32 | 32
units on a scale | 1.5 (0.88) | 1.4 (0.84)

ADVERSE EVENTS:
Arm/Group | Juvederm Ultra Injectable Gel With Lidocaine | Restylane
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 2/32 | 8/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Juvederm Ultra Injectable Gel With Lidocaine (N=32) | Restylane (N=32)
Injection site swelling (General disorders) | 1 (1) | 3 (3)
Injection site pain (General disorders) | 1 (1) | 3 (3)
Injection site induration (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.